CLINICAL TRIAL: NCT02623062
Title: A Multi-centred, Randomised, Double-blind, Two Arms, Parallel Group, Placebo-controlled Study to Assess the Effect of Compound Sodium Alginate Oral Suspension Sachet in Patients With Reflux Disease
Brief Title: Compound Sodium Alginate Oral Suspension Sachet Symptomatic Relief Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GA1217
Record Dates: First submitted 2015-11-30; First posted 2015-12-07 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Gastro-esophageal Reflux Disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Compound Sodium Alginate Oral Suspension sachets (Active Comparator): Each patient will be instructed to take Compound Sodium Alginate Oral Suspension sachet or matching placebo as a 2x10ml sachets four times daily regimen. Prior to dosing, all patients will be instructed by the Investigator on how they will take the medication. Patients will be instructed to start taking their medication the day after their randomisation visit (Day 1) for seven days (20ml taken four times a day: 30 minutes after breakfast, 30 minutes after lunch, 30 minutes after dinner and immediately before lying down for bed. Shake well before use).
  Interventions: Drug: Compound Sodium Alginate Oral Suspension sachet
- Matching placebo sachets (Placebo Comparator): Each patient will be instructed to take Compound Sodium Alginate Oral Suspension sachet or matching placebo as a 2x10ml sachets four times daily regimen. Prior to dosing, all patients will be instructed by the Investigator on how they will take the medication. Patients will be instructed to start taking their medication the day after their randomisation visit (Day 1) for seven days (20ml taken four times a day: 30 minutes after breakfast, 30 minutes after lunch, 30 minutes after dinner and immediately before lying down for bed. Shake well before use).
  Interventions: Drug: Matched placebo

INTERVENTIONS:
Drug: Compound Sodium Alginate Oral Suspension sachet — Contents of 2 sachets taken four times daily for 7 days
  Other Names: Gaviscon sachets
  Arms: Compound Sodium Alginate Oral Suspension sachets
Drug: Matched placebo — Contents of 2 sachets taken four times daily for 7 days
  Other Names: Placebo
  Arms: Matching placebo sachets

SUMMARY:
This study is being conducted in China to provide evidence for inclusion in applications to competent authorities that the Compound Sodium Alginate Oral Suspension sachet is effective in managing the symptoms of heartburn and acid regurgitation in patients with gastro-esophageal reflux disease (GERD).

DETAILED DESCRIPTION:
This is a multi-centre, randomised, double blind, two arm, parallel group, placebo-controlled clinical trial in patients with moderate to severe and frequent GERD symptoms. After signing a written informed consent, patients will undergo a screening period of up to 7 days. Patients who satisfy the study entry requirements within 7 days of consent, will be randomised to receive either Compound Sodium Alginate Oral Suspension sachets (20ml four times daily) or matching placebo sachets (20ml four times daily),for a 7- day treatment period. At the beginning and end of the treatment period, patients will be required to complete the Reflux Disease Questionnaire (RDQ).

In addition, at the end of the 7 (-1 day to +2 days) day treatment period, patients will be required to complete the Overall Treatment Evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis: Current evidence of symptomatic GERD/NERD that comply with the Montreal definition of GERD/Nonerosive Esophageal Reflux Disease (NERD). GERD is a condition which develops when the reflux of stomach contents causes troublesome symptoms and/or complications. The concept of NERD is preserved in the typical reflux syndrome without esophageal injury, while reflux esophagitis falls under the category of esophageal syndromes with esophageal injury.
* GERD status: patients will be recruited by the Investigator from out-patient clinics, hospital database or those who respond to the advertising. Patients must have a GERD history of frequent episodes of GERD-related symptoms during the last 3 months, and must have had troublesome heartburn and/or regurgitation of at least moderate intensity on at least 4 days during the week before the start of screening.
* Patients must be sufficiently literate to be able to complete the RDQ unaided.

Exclusion Criteria:

* Patients who have a history of drug, solvent or alcohol abuse (weekly alcohol intake ≥ 140g).
* Patients who have suffered cardiac chest pain within the last year.
* Patients who have suffered a recent, significant unexplained weight loss of more than 6 kg in the last 6 months.
* Female patients of childbearing potential who, for the duration of the study, are either unwilling or unable to take adequate contraceptive precautions or are unwilling to be sexually abstinent.
* Pregnancy or lactating mother.
* Patients with a history and/or symptom profile suggestive of the following: any other gastrointestinal (GI) disease (e.g. gastric or duodenal erosions and polyps larger than 0.5 cm), erosive GERD (Los Angeles [LA] classification grades C-D), Barrett's esophagus, peptic ulcer and/or ulcer complications, Zollinger-Ellison syndrome, gastric carcinoma, pyloric stenosis, oesophageal or gastric surgery, intestinal obstruction, current pernicious anaemia, indication for H-pylori eradication, hiatal hernias greater than 3 cm, known gastro-intestinal bleeding (hematochezia or hematemesis) within the last 3 months, and severe diseases of other major body systems.
* Patients who have taken anti-cholinesterase drugs, traditional Chinese medicines for treating gastrointestinal disease, Ulcermin or misoprostol preparations within 7 days prior to screening or throughout the study.
* Patients who have taken Proton Pump Inhibitors (PPIs) during the 10 days prior to screening, prokinetics or H2 antagonists during the 5 days prior to screening, or systemic glucocorticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs except low dose aspirin given for cardioprotection) on more than 3 consecutive days during the last 28 days prior to screening or PPI-based triple or quadruple therapy for eradication of H-pylori during the last 28 days prior to screening and throughout the study.
* Patients who have taken any antacids within 24 hours before randomisation (Visit 2) and are unwilling or unable to withhold from taking them for the duration of the study.
* Patients taking mucous membrane protection drugs or motility stimulants within the 5 days prior to screening and are unwilling or unable to withhold from taking them for the duration of the study.
* Patients with difficulty in swallowing.
* Patients with known hypophosphataemia, phenylketonuria or hypercalcaemia.
* Patients with severe constipation, or history of intestinal obstruction.
* In the opinion of the Investigator, patients with insufficient heart or kidney function and patients who require a low sodium diet.
* Patients with any co-existing condition which, in the opinion of the Investigator, would be likely to compromise patient safety or interfere with assessment of efficacy.
* Patients with any clinically significant abnormal laboratory values.
* Patients with severe/impaired renal function or insufficiency.
* Any previous history of allergy or known intolerance to any of the formulation constituents.
* Relevant clinically significant abnormalities in the physical examination, ECG and safety analysis.
* Previously randomised into the study.
* Employee at study site.
* Partner or first-degree relative (e.g. parents, siblings or children) of the Investigator.
* Participation in a clinical study in the previous 6 months.
* Unable in the opinion of the Investigator to comply fully with the study requirements.
* Patients taking or requiring to take macrolide antibiotics, such as erythromycin, azithromycin, from the day before screening
* Patients who failed screening will not be allowed to re-enter the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2013-12; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in GERD dimension of RDQ | 0 and 7 days
  Change from day 0 in the GERD dimension (heartburn and regurgitation combined) from the RDQ symptom scores after a 7-day treatment period

SECONDARY OUTCOMES:
Change in symptom score for each dimension of the RDQ separately | 0 and 7 days
  Change from day 0 in symptom score for each dimension of the RDQ separately (heartburn and regurgitation)
Change in frequency of each symptom separately (heartburn and regurgitation) from RDQ assessment | 0 and 7 days
  Change from day 0 in frequency of each symptom separately (heartburn and regurgitation) from RDQ assessment.
Change in intensity of each symptom separately (heartburn and regurgitation) from RDQ assessment | 0 and 7 days
  Change from day 0 in intensity of each symptom separately (heartburn and regurgitation) from RDQ assessment
Change in symptoms using the Overall Treatment Evaluation (OTE) | 0 and 7 days
  Rating of change in symptoms using the Overall Treatment Evaluation (OTE)

CONTACTS AND LOCATIONS:
Overall Officials: MinHu Chen, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affilated Hospital Sun Yat-Sen University, Guangzhou, Guangdong, China